CLINICAL TRIAL: NCT03710954
Title: Application and Comparison of Fuzzy Scale for the Evaluation of Pain Skeletal Muscle With the Numerical Pain Scale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cruzeiro do Sul (Other)
Responsible Party: Principal Investigator, Leandro Lazzareschi, PhD, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17258413.0.0000.5497
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pain
Keywords: Evaluation of pain; Fuzzy systems theory
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): All the volunteers were evaluated through numerical evaluation of pain that assumes a subjective condition, the researcher showed the numerical scale of pain, being 0 without pain, 1 to 4 mild pain, 5 moderate pain, 6 to 9 severe pain and 10 worse pain possible pain, which was interpreted by the volunteer. In the Fuzzy Pain Scale, the evaluation of the range of motion was done where the evaluator used the goniometer (plastic instrument that verifies the angulation of the joint movement) and supplied the Fuzzy system with these data.
  Interventions: Diagnostic Test: Experimental Group

INTERVENTIONS:
Diagnostic Test: Experimental Group — All volunteers were evaluated by numerical pain scale and Fuzzy scale. This procedure was performed to compare the efficacy of the Fuzzy Scale demonstrating greater accuracy of quantification of skeletal muscle pain

SUMMARY:
This study aimed to analyze the stratification of pain levels through a mathematical model built using the diffuse joint theory and to investigate the relationship between range of motion and pain related aspects.

DETAILED DESCRIPTION:
The incidence of pain is due to traumatic actions, surgical interventions, new habits of life, increased longevity of the individuals and the reduction of the tolerance of the suffering by the man. Musculoskeletal pain is more evident in adult individuals, being the main cause of chronic pain throughout society, generating an impact on the quality of life, interfering in the daily activity of 30 to 50% of the patients. Pain measurement can be divided into four levels, which include the nominal, the ordinal, the interval and the ratio, with both one-dimensional and multidimensional versions. In the health area, diagnosis and treatment of diseases involve various levels of imprecision and uncertainties. A single disease or symptom may manifest totally differently in different patients and with varying degrees of severity. These effects usually generate many uncertainties and inaccuracies affecting the interpretations of the exams and the diagnosis, as well as the treatment. Fuzzy Systems Theory, also known as nebulous logic, is used to interpret the approximate mode of human reasoning, to take it to a numerical format and to obtain answers in an environment of uncertainties that serve as a subsidy to decision-making . A Fuzzy system based on Fuzzy logic. It can also be considered as a kind of expert, knowledge-based system. The development of the proposed Fuzzy Scale for Skeletal Muscle Pain Evaluation used the Mamdani method that allowed the representation of specialist knowledge (s) to construct the rule base. The construction of this system was based on the numerical scale of pain adopted and spread worldwide, and on the range of motion represented by the action of the muscles and articular components of the human body. The diffuse model proposed by the Fuzzy Scale for Muscle Skeletal Pain Evaluation uses 25 rules using binary XOR logic. For the volunteer tests, the proposed model was a non-randomized single intervention transverse study to analyze and compare the model of diffuse pain evaluation with the numerical pain scale performed with 535 volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Included in this study were male and female subjects
* Age between 18 and 90 years
* With complaint of skeletal muscle pain
* Do not present cognitive deficit that makes the study impossible

Exclusion Criteria:

* Individuals who did not agree to participate in the study
* Volunteers with decreased range of motion
* Volunteers without complaint of skeletal muscle pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 535 individuals with complaint of skeletal muscle pain
Enrollment: 535 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Numerical scale of pain | 10 minutes
  Patients across this scale quantified their pain between 0 without pain, 1 to 4 mild pain, 5 moderate pain, 6 to 9 severe pain and 10 worst possible pain

SECONDARY OUTCOMES:
Fuzzy Pain Scale | 10 minutes
  The evaluation of the range of motion was done by an evaluator who used a goniometer (plastic instrument that verifies the angulation of joint movement) according to: Spine-cervical Flexion: 0-65°; Cervical extension: 0-50°; Shoulder-horizontal Adduction: 0-40°; Internal rotation: 0-90°; External rotation: 0-90 °; Flexion: 0-145°; Extension: 145-0°; Elbow: Pronation: 0-90°; Supination: 0-90°; Flexion: 0-90°; Fist-extension: 0-75°; Radial deviation: 0-25ø; Ulnar deviation: 0-45°; Flexion: 0-95 °; Extension: 0-35 °; Lumbar spine-lateral flex: 0-40 °; Trunk rotation: 0-35 °; Flexion (knee flexion): 0-125°; Flexion (knee extended): 0-90°; Extension: 0-10°; Hip-external rotation: 0-45°; Abduction: 0-45°; Adduction: 0-15°; Flexion: 0-140°; Knee-Bending: 0-140°; Ankle-Dorsiflexion: 0-20°; Plant flexion: 0-45°. Supplying the Fuzzy Pain Analysis System.

IPD SHARING:
Plan to Share IPD: No